# An Exploratory Open-Label Potency and Precision Investigation of a Relational Agent Intervention

NCT06240091

March 18, 2024



Protocol Number: W-DISC-002

NCT Number: NCT06240091

Date 18/MAR/2024

#### W-DISC-002

An Exploratory Open-Label Potency and Precision Investigation of a Relational Agent Intervention

Document Type: Clinical Trial Protocol

Clinical Trial Phase: Phase I/II

Version Number: 1.1

Property of Woebot Health
Confidential

May not be used, divulged, published, or otherwise disclosed without the consent of Woebot Health

# **CLINICAL STUDY PROTOCOL**

# An Exploratory Open-Label Potency and Precision Investigation of a Relational Agent Intervention

| Protocol Number | W-DISC-002 |
|---|---|
| Investigational Product | DISC-MA |
| Sponsor | Woebot Health 535 Mission Street, 14th Floor San Francisco, CA 94105 |
| Principal Investigator | Tim Campellone, PhD tim_campellone@woebothealth.com |
| Version | 1.1 |
| Date | 18/MAR/2024 |

This study will be performed in compliance with the principles of Good Clinical Practice.

# **Protocol Version and Amendment Tracking**

| Version | Date | Brief Summary of Changes |
|---|---|---|
| 1.0 | 21/DEC/2023 | Original Protocol |
| 1.1 | 18/MAR/2024 | Updated administration timeline for the NIH Toolbox Social Relationship scales (i.e., removed Week 2 assessment point), added in details for an optional post trial user experience interview, and added clarifying language around safety monitoring procedures. |

# **Confidentiality Statement**

The information in this protocol is confidential and proprietary information of Woebot Health. It is provided to you as a site, Investigator or consultant for review by you, your staff, and other applicable regulatory bodies. Acceptance of this document constitutes agreement that you will not disclose the information contained herein to others without written authorization from the Sponsor or in a way that is inconsistent with contractual language.

# **Protocol Signature Page | Sponsor**

This protocol has been reviewed and approved by the representative(s) listed below. Any modification of the protocol must be agreed upon by the Sponsor and the investigator and must be documented in writing.

| ebot Health Representative(s): | |
|-----------------------------------------------|------------------|
| [Principal Investigator or Sponsor Signature] | [Signatory Date] |
| [Name and Title of Signatory] | |

# **Protocol Signature Page | Principal Investigator**

I have read this protocol, which has been agreed by Woebot Health, and given approval/favorable opinion by the institutional review board, and I agree that it contains all necessary details for my staff and I to conduct this study as described. I will provide copies of the protocol and any amendments to all study personnel under my supervision and provide access to all information provided by Woebot Health or their specified designees. I will discuss the material with the study personnel to ensure that they are fully informed about the study.

I understand that information contained in or pertaining to this protocol is confidential and should not be disclosed, other than to those directly involved in the execution or the ethical review of the study, without written authorization from Woebot Health. It is, however, permissible to provide information to a participant in order to obtain consent.

I agree to conduct this study according to this protocol and to comply with its requirements, participant to ethical and safety considerations and guidelines, and to conduct the study in accordance with the Declaration of Helsinki, International Council for Harmonisation guidelines on Good Clinical Practice, and applicable regional regulatory requirements.

I agree to comply with the procedures described for data recording and reporting and to permit monitoring and auditing by Woebot Health and inspection by the appropriate regulatory authorities.

I agree to make my participants' study records available to Woebot Health personnel, their representatives, and relevant regulatory authorities in order to verify data that I have entered in the case report forms. I will retain the study-related essential documents until Woebot Health indicates that they are no longer needed. I am aware of my responsibilities as an investigator as provided by Woebot Health.

I understand that Woebot Health may decide to suspend or prematurely terminate the study at any time for whatever reason; such a decision will be communicated to me in writing. Conversely, should I decide to withdraw from execution of the study, I will communicate my intention immediately in writing to Woebot Health.

| [Principal Investigator Signature] | [Date] |
|------------------------------------|--------|
| | [Site] |

# **Protocol Synopsis**

| Protocol Number: | W-DISC-002 |
|---|---|
| Full Title: | An Exploratory Open-Label Potency and Precision Investigation of a Relational Agent Intervention |
| Abbreviated Title: | PAPI: Potency and Precision Investigation |
| Sponsor: | Woebot Health |
| Study Type: | Product learning |
| Number of Participants: | 200 |
| Number of Sites: | 1 |
| Study Objective: | The overarching goal of this study is to establish initial proof of mechanism for precision interventions in an adult population. |
| Primary Aim and Endpoint: | Aim: Describe therapeutic alliance with Woebot at week 1 and week 4 of the intervention. Endpoints: Working Alliance Inventory (WAI) total score at week 1 and WAI total score at week 4. |
| Secondary Aims and Endpoints: | N/A |

W-DISC-002 18/MAR/2024

Version 1.1



| Study Design: | Single arm pilot study |
|---|---|
| Study Duration: | 4 week intervention period |
| Target Population: | Adults between the ages of 18 and 75 years experiencing at least mild depression or anxiety symptoms. |
| Key Inclusion Criteria: | <ol> <li>Adults 18 - 75</li> <li>Has regular access to a smartphone (Android or iOS smartphone with a recent supported operating system) with reliable WiFi access or sufficient data to engage with assigned study arm for the duration of the study</li> <li>Available and committed to engage with the program and complete assessments for study duration</li> <li>Able to read and write in English</li> <li>U.S. resident</li> <li>PHQ-8 &gt; 4 and/or GAD-7 &gt; 4, assessed at Screening/Baseline</li> </ol> |
| Key Exclusion Criteria: | <ol> <li>Current suicidal ideation with a plan and/or intent or a suicide attempt within the past 12 months</li> <li>Previous Woebot use</li> <li>Involuntary inpatient psychiatric hospitalization any time within the past 30 days</li> <li>Lifetime diagnosis of bipolar disorder</li> <li>Lifetime diagnosis of a psychotic disorder</li> </ol> |
| Study Condition: | DISC-MA |

Version 1.1

18/MAR/2024

| Test Device: | DISC-MA |
|---|---|
| Control Device: | N/A |
| Statistical Methods: | Descriptive statistics will be reported for study measures. Summary reports will be presented for all time periods independently. Bivariate analyses will use chi-squared tests, Fisher exact test, t-tests, one-way ANOVA, Person's correlation, and Spearman's correlation, where applicable. No hypothesis testing will be completed, and only effect sizes and 95% confidence intervals will be provided where applicable. For departures from normality, the appropriate non-parametric method will be applied. |
| Protocol Version and Date: | 1.1 (18 /MAR /2024 ) |
| Keywords: | digital mental health intervention, chatbot, conversational agent, relational agent, natural language processing, artificial intelligence |

Woebot Health Version 1.1 18/MAR/2024

# W-DISC-002

**Table of Contents** 

| Table 1. Schedule of Events | 13 |
|-----------------------------------------------|----|
| 1. Introduction | 14 |
| 1.1 Background | 14 |
| 1.2 Study Rationale | 14 |
| 1.3 Investigational Device | 14 |
| 2. Objectives | 15 |
| 2.1 Primary Aim | 15 |
| 3. Study Design | 16 |
| 3.1 Description of Trial Design | 16 |
| Figure 2: Participant Journey Flowchart | 17 |
| 3.2 Rationale for Trial Design | 17 |
| 4. Trial Intervention | 17 |
| 4.1 Study Condition | 17 |
| 4.3 Trial Intervention Compliance | 18 |
| 5. Study Population | 18 |
| 5.1 Selection of Study Population | 19 |
| 5.1.1 Inclusion Criteria | 19 |
| 5.1.2 Exclusion Criteria | 19 |
| 5.2 Screen Failures | 19 |
| 5.3 Withdrawal of Participants from the Study | 20 |
| 6. Study Assessments and Procedures | 20 |
| 6.1 Pre-Screening Procedures | 21 |
| 6.2 Screening Assessments and Procedures | 21 |
| 6.2.1 Identity Verification Call | 21 |
| 6.2.2 Demographic Questions | 21 |
| 6.2.3 Medical History | 21 |
| Prior and Concomitant Medication and Therapy | 21 |
| Psychiatric History | 21 |
| 6.3 Primary Endpoint | 21 |
| Working Alliance Inventory (WAI-SR) | 21 |

W-DISC-002

29

30

30

30

| | <u> </u> |
|------------------------------------------------------|----------|
| | <u> </u> |
| | <u> </u> |
| | <u> </u> |
| | <u> </u> |
| | <u> </u> |
| | <u> </u> |
| | <b>_</b> |
| 7. Charle Characine Bules | 24 |
| 7. Study Stopping Rules | 24 |
| 7.1 Early Study Termination | 24 |
| 8. Data and Safety Monitoring | 25 |
| 8.1 Risk and Benefit Assessment | 25 |
| 8.1.1 Risks | 25 |
| 8.1.2 Procedures for minimizing risk | 25 |
| Misunderstanding the Capabilities of the Application | 25 |
| Data Breach | 25 |
| Potential Upset due to Study Procedures | 25 |
| 8.1.3 Benefits | 26 |
| 8.2 Adverse Events | 26 |
| 8.2.1 Definitions | 26 |
| 8.2.2 Previously Noted Adverse Device Effects | 28 |
| 8.3 Assessment of Adverse Events | 28 |
| 8.3.1 Time Frame | 28 |
| 8.3.2 AE Severity | 28 |
| 8.3.3 AE Causality | 29 |
| 8.3.3 AE Outcomes | 29 |
| 8.4 Documenting and Reporting AE and SAEs | 29 |
| 8.5 Safety Monitoring | 29 |

CONFIDENTIAL 11

8.5.1 Safety Procedures At Screening

8.5.3 Safety Event Solicited Self-Report Survey

8.5.4 Language Detection Protocol (LDP)

8.5.2 Unscheduled Visits

| Woebot Health | Version 1.1 |
|------------------------------------------------------|-------------|
| W-DISC-002 | 18/MAR/2024 |
| 8.6 Safety Assessment Committee (SAC) | 32 |
| 8.6.1 Risk and Quality Tolerance Limits | 33 |
| 8.7 Quality Control and Quality Assurance | 33 |
| 9. Statistical Analysis | 33 |
| 9.1 General Methodology | 33 |
| 9.2 Analysis Sets | 33 |
| 9.3 Sample Size Determination | 34 |
| 10. Statistical Methods | 34 |
| 10.1 Primary Endpoint | 34 |
| 10.1.1 Aim | 34 |
| 10.1.2 Hypothesis | 34 |
| 10.1.3 Endpoints | 34 |
| 10.1.4 Analysis Plan | 34 |
| 10.3 Safety Endpoints | 35 |
| 10.3.1 Aims and Endpoints | 35 |
| 10.3.2 Analysis of Safety | 35 |
| 10.4 Demographic and Baseline Characteristics | 35 |
| 10.5 Handling of Missing Values | 35 |
| 11. Ethics and Responsibilities | 36 |
| 11.1 Good Clinical Practice | 36 |
| 11.2 Institutional Review Board | 36 |
| 11.3 Informed Consent | 36 |
| 12. Records Management | 37 |
| 12.1 Source Documentation | 37 |
| 12.2 Case Report Form Completion and Data Management | 38 |
| 12.3 Study Files and Record Retention | 38 |
| 13. Auditing and Monitoring | 39 |
| 13.1 Protocol Adherence and Deviations | 39 |
| 14. Amendments | 40 |
| 15. Study Start and Termination | 40 |
| 16. Confidentiality | 40 |
| 17 References | //2 |

W-DISC-002 18/MAR/2024

**Table 1. Schedule of Events** 

| | Screening Period Intervention Period | | | |
|---|---|---|---|---|
| Visit Weeks/Days | Screening / Baseline | Week 1 | Week 2 | Week 4 |
| | Day -14 to Day 1 | Day 7 (+6) | Day 14 (+6) | Day 28 (+6) |
| Informed Consent (asynchronous e-Consent via Citrus) | х | | | |
| Participant Identity Verification <sup>a</sup> | Х | | | |
| Eligibility Confirmation (inc/exc) <sup>b</sup> | Х | | | |
| Demographics <sup>b</sup> | Х | | | |
| Medical History Prior & Concomitant<br>Medications/Therapy <sup>b</sup> | Х | | | |
| Medical History Psychiatric History b | Х | | | |
| The Accountable Health Communities Health-Related Social Needs Screening Tool b | Х | | | |
| | | | | _ |
| App Download / Registration <sup>c</sup> | X | | | |
| Working Alliance Inventory (WAI-SR) <sup>b</sup> | | Х | | Х |
| Safety Survey <sup>b</sup> | | | X | х |
| Assessment of AE/SAEs | | x | | |
| Enactment <sup>c</sup> | | X | | |
| App Engagement Metrics <sup>c</sup> | | | X | |
| Termination of App Access <sup>c</sup> | | | | Х |
| Estimated Time to Complete | 45 minutes | 15 minutes | 30 minutes | 30 minutes |

<sup>&</sup>lt;sup>a</sup> Live video call with Lindus Health trial team <sup>b</sup> Self-report through Citrus platform <sup>c</sup> Study app

Participants will have up to two weeks from the time of providing informed consent to complete all screening and baseline tasks including registering for the study application. Participants will be considered a screen fail and removed from the study for failing to register for the app by Day 3.

#### 1. Introduction

#### 1.1 Background

Precision medicine is defined by the Food and Drug Administration as "...to target the right treatments to the right patients at the right time". In the context of mental health, the goal of a precision medicine approach is to use the various tools and data to develop more effective and safe treatments<sup>2</sup>. Digital mental health interventions are uniquely positioned to create and deliver precision interventions that follow this FDA definition by being able to deliver in a standardized way fit for purpose interventions that target mechanisms for specific users at specific moments of the user journey.

#### 1.2 Study Rationale

The overarching goal of this study is to inform the development of precision interventions within the Woebot for Mood and Anxiety investigational product. This study will provide initial learning on the current implementation of precision interventions and generate data and hypotheses to inform the exploration of future interventions by identifying mechanisms and moments in the user journey to target.

#### 1.3 Investigational Device

| DISC-MA is a discovery version (3.2) of the investigational product Woebot for Mood and Anxiety and is a non-prescription digital software device, accessible via iOS and Android smartphone operating systems. |
|---|

W-DISC-002 18/MAR/2024



# 2. Objectives

# 2.1 Primary Aim

- Describe therapeutic alliance with Woebot at week 1 and week 4 of the intervention.
- Primary Endpoints:
  - Working Alliance Inventory (WAI) total score at week 1 and WAI total score at week 4.



Woebot Health Version 1.1



# 3. Study Design

#### 3.1 Description of Trial Design

This study is a single arm pilot trial aimed at exploring and informing precision interventions within the Woebot for Mood and Anxiety investigational device. Study participation is up to 7 weeks in total, including a 2 week screening/baseline phase, followed by a 4 week active intervention phase, and 1 week to complete the final study survey.

Participants will be recruited and enrolled into the study by Lindus Health. All remaining data collection and study monitoring will be managed through the Citrus decentralized trial platform managed by Lindus Health and by designated Woebot Health study personnel.

Self-report survey assessments will be administered to all participants at Screening/Baseline, Week 1, Week 2, and Week 4. Members of the study team may contact participants through the Citrus platform via phone/sms and/or email to remind participants to complete study activities.

**Figure 2: Participant Journey Flowchart** 



# 3.2 Rationale for Trial Design

This trial design will allow for characterization of participants at baseline in order to better understand and generate hypotheses about how these characteristics interact with patterns of engagement within the Woebot for Mood and Anxiety investigational product.

## 4. Trial Intervention

# **4.1 Study Condition**

All participants will have access to the same trial intervention, DISC-MA, for 4 weeks. The trial intervention will be accessed through a mobile app and will be made available exclusively for study participants through unique access codes.



# **4.3 Trial Intervention Compliance**

Participants will be removed from the study and considered a "screen failure" for failing to register for the app by Day 3. Trial intervention compliance will not be monitored during the live trial and participants will not be withdrawn for not regularly engaging with their assigned treatment. Instead, intervention compliance will be assessed post study during analysis. Compliance may be defined as opening the app at least once per week for a minimum of 50% of weeks (2 of 4) during the intervention period.



## **5. Study Population**

Participants will be recruited through the Lindus Health CitrusRecruit network which utilizes a combination of participant sources including but not limited to existing patient databases, primary care networks, and targeted social media campaigns. Those interested in participating will be invited to complete a survey to confirm they meet the pre-screening criteria and be presented with the opportunity to independently review and electronically sign the study consent form. Upon signing the consent form, participants will be asked to schedule a video call during which a designated member of the Lindus Health trial team will verify the participants identity. After successful completion of the verification call, participants will be provided with a secure link to complete the screening/baseline survey. In order to further assess eligibility, participants will be asked questions about their medical history including self-report of (1) any involuntary inpatient psychiatric hospitalizations within the past 30 days, (2) a lifetime diagnosis of bipolar disorder, (3) a life time diagnosis of a psychotic disorder, and

(4) current suicidal ideation with plan and/or intent or an attempt in the past 12 months. People who do not meet study criteria based on these additional exclusionary criteria will be notified that they may benefit from a level of care beyond the scope of the study and that if they feel they are in need of immediate medical care they should contact 911 or go to their nearest emergency room and reach out to someone they trust and that can help them stay safe. Additional resources will also be provided electronically. If a participant endorses presence of <u>current</u> suicidal plan and/or intent, the study PI will attempt to follow-up with the participant (up to three times). See Section 8.5.1 of this protocol for more details.

#### **5.1 Selection of Study Population**

The study aims to enroll approximately 200 adults between the ages of 18 and 75 years experiencing at least mild depression or anxiety symptoms into the study. An enrolled participant is defined as a participant that meets all eligibility criteria as described below and registers in the app by Day 3 of the study.

#### 5.1.1 Inclusion Criteria

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

- 1. Adults between the ages of 18 and 75 years
- 2. Own or have regular access to a smartphone with a recent operating system installed (Android: 0S 8.0 or higher, Apple: iOS 13.0 or higher) with reliable Wi-Fi access or sufficient data plan to engage with assigned treatment condition for the duration of the study
- 3. Available and committed to engage with the program and complete assessments for a 4-week duration
- 4. Able to read and write in English
- 5. U.S. resident
- 6. PHQ-8 > 4 and/or GAD-7 > 4, assessed at screening/baseline

#### 5.1.2 Exclusion Criteria

An individual who meets any of the following criteria will be excluded from participation in this study:

- 1. Current suicidal ideation with a plan and/or intent or a suicide attempt within the past 12 months
- 2. Previous Woebot use
- 3. Involuntary inpatient psychiatric hospitalization any time within the past 30 days
- 4. Lifetime diagnosis of bipolar disorder
- 5. Lifetime diagnosis of a psychotic disorder

#### **5.2 Screen Failures**

Participants who sign study consent and (1) do not meet inclusion/exclusion criteria or (2) fail to register in the app by Day 3, will be considered a Screen Failure. Participants will be notified that they did not meet eligibility criteria and provided with a set of resources. Re-screens will not be permitted in this study. De-identified participant ID numbers assigned to participants who screen fail will not be reused.

## 5.3 Withdrawal of Participants from the Study

If a participant decides to withdraw consent from the study, they will be removed from future study activities and any data collected before withdrawal may be retained and used in study analyses. In addition, a participant may be withdrawn by the investigator if the participant violates the study plan, or for administrative and/or other safety reasons.

Discontinuation of study treatment for a participant occurs when study treatment is stopped earlier than the protocol planned duration and can be initiated by either the participant or the investigator. The investigator must discontinue study treatment for a given participant if he/she believes that continuation would negatively impact the participant's well-being. Involvement in the study is strictly voluntary. Participants have the right to withdraw from the study at any time for any reason, without any reprisal.

Participants should be discontinued from the study if any of the following occur:

- 1. It is discovered that the participant shared app images/screenshots publicly
- 2. The participant withdraws consent to participate in the study
- 3. The participant develops an illness that would interfere with their continued participation in the study
- 4. The participant has an SAE rated as Grade 3 (severe) or higher (see Section 8.3.2)
- 5. The participant is noncompliant with treatment schedule, study procedures, in the opinion of the investigator and per the protocol, where applicable
- 6. The PI, Sponsor, IRB, or regulatory agency requests withdrawal of the participant
- 7. Any other reason relating to the participant's safety or integrity of the study data as determined by the Safety Assessment Committee (SAC)

Participants who withdraw or are withdrawn from the study may be replaced. Participants who withdraw or are withdrawn from the study cannot subsequently rejoin the study.

If a participant withdraws or is withdrawn from the study for reasons related to safety, the study Sponsor-Investigator and SAC will be informed immediately.

If the participant withdraws consent for disclosure of further information, the Sponsor-Investigator may retain and continue to use any collected data before such a withdrawal of consent.

Although a participant is not obliged to give a reason for withdrawing from a study, the investigator should make a reasonable effort to ascertain the reason, while fully respecting the participant's rights.

#### 6. Study Assessments and Procedures

All assessments, and their corresponding administration points, are listed in Table 1.

#### **6.1 Pre-Screening Procedures**

Participants will have the opportunity to learn about the study through digital recruitment efforts. Interested participants will complete a pre-screening survey to determine preliminary eligibility ahead of consent. Eligible participants at this stage will then proceed to review and sign the eICF.

#### **6.2 Screening Assessments and Procedures**

#### **6.2.1 Identity Verification Call**

After passing pre-screening criteria and signing the study eICF, participants will be asked to schedule an identity verification video call with a member of the Lindus Health study team. During this call the designated member of the study team will ask the participant to verify their identity (e.g., show a government issued ID) as well as confirm their contact information and DOB.

#### **6.2.2 Demographic Questions**

In an effort to ensure equitable access and representation as well as assess clinical efficacy in diverse populations, Woebot Health has researched current best practices and language around demographic data collection, and developed a health equity demographic battery. The demographic battery consists of age, biological sex, gender identity, sexual orientation, race, ethnicity, education, marital status, employment status, living situation, able bodiedness, physical health conditions, and health insurance status.

#### **6.2.3 Medical History**

#### **Prior and Concomitant Medication and Therapy**

Participants will be asked to complete questions evaluating whether they are currently seeing a mental health professional (i.e., therapist, social worker), whether they are currently taking any psychotropic medications, as well as satisfaction with concurrent mental health treatment.

#### **Psychiatric History**

Participants will be asked to complete questions about their history of diagnosed mental health disorders including self-report of a lifetime diagnosis of bipolar disorder and/or a psychotic disorder as well as whether they have current suicidal ideations with plan and/or intent or if they have had a suicide attempt in the past 12 months. Participants will also be asked to endorse whether they have experienced any involuntary inpatient psychiatric hospitalizations within the past 30 days.

#### **6.3 Primary Endpoint**

#### Working Alliance Inventory (WAI-SR)

The WAI-SR<sup>5</sup> is a measure of therapeutic bond and consists of a composite score and three subscales; Bond, Goal, and Task. Bond measures the strength of the therapeutic relationship between the client and therapist. Goal measures agreement on the goal of the overall therapeutic program between the client and therapist. Task measures agreement between the client and therapist, regarding the specific activities needed for a therapeutic change to occur such as doing an exercise to ameliorate a specific

W-DISC-002 18/MAR/2024

symptom3. The present study utilized the validated 12-item Short Revised version (WAI-SR) with minor changes to language, replacing "therapist" with the name of the assigned treatment group.



Woebot Health Version 1.1



# 7. Study Stopping Rules

Study procedures will be stopped if the Sponsor-Investigator, in discussion with the SAC and/or IRB as applicable, determines that the number and/or severity of AEs justify putting the study on hold.

The study may resume following the safety review, if the Sponsor-Investigator agrees it is safe to proceed.

The Sponsor-Investigator may initiate study closure at any time, provided there is reasonable cause and sufficient notice is given in advance of the intended termination.

# 7.1 Early Study Termination

The study can be terminated by the Sponsor-Investigator at any time. Reasons for early termination include:

- Study recruitment or retention is too low for the study to provide meaningful results
- Unanticipated, significant, or unacceptable safety risk to participants enrolled in the study
- Decision based on recommendations from Sponsor-Investigator and SAC after review of safety and efficacy data
- Discontinuation of study if Sponsor-Investigator, in collaboration with study team members and SAC, determine from planned analyses that the app is not efficacious or if there are safety concerns.

In making the decision to terminate, the Sponsor-Investigator and SAC will always consider the participants' welfare and safety. Should early termination be necessary, participants must be contacted as soon as possible to conduct EOS assessments, if willing, and treated as a prematurely withdrawn participant. Additional procedures may be provided to ensure that adequate consideration is given to the protection of the participant's interests. The Sponsor-Investigator will be responsible for informing IRB of the early termination of the trial.

# 8. Data and Safety Monitoring

#### 8.1 Risk and Benefit Assessment

#### 8.1.1 Risks to Participants

Given that the research aims to enroll participants into a low-risk intervention, we do not anticipate that participation in the study will be associated with elevated risk.

The overall

evaluation of risk is that it is low.

## **8.1.2 Procedures for minimizing risk**

#### Misunderstanding the Capabilities of the Application

DISC-MA is not intended to be a crisis service, however there is the potential that participants may misunderstand the limitations of the app. To mitigate this risk, the study will provide clear information on the capabilities of the app, intended use, and limitations of the app at consent, treatment assignment, and key points throughout. Resources are also accessible within the app as well and will be sent to the participant in the event that they are requested.

#### Data Breach

All study data are gathered on either a HIPAA-compliant web platform that resides behind Woebot Health security firewalls or via HIPAA-compliant online platforms, thus actual risk from data breach for study data is low. Research material obtained from human subjects will include self-report questionnaires and conversations and engagement data within the mobile app. All data obtained via Woebot will be encrypted and stored on Amazon Web Services (AWS) and/or Google Cloud Platform; Woebot Health data gathering and storage procedures are compliant with both HIPAA and the European Union's General Data Protection Regulation. Only members of the research team will have access to identifiable study data. De-identified data will be accessible to the product development team (designers, user researchers, and product managers) as well as the research team.

#### Potential Upset due to Study Procedures

Foreseeable risks to participants include the possibility that some assessment questions and/or treatment procedures may be upsetting to participants. Experience with similar populations has indicated that the risk of emotional upset during the assessments is low and if it occurred, the upset would likely be temporary and not be serious in nature. Such risks will be minimized by the thoughtful selection of questionnaires. Participants will also be informed that they may withdraw from the study at any time and if requested, appropriate resources will be provided.

There is also a potential risk for upset upon discontinued access to the study intervention at end of treatment/study (Week 4). Participants are informed during the consent process and are reminded at onboarding of how long they will have access to the intervention for. Return to care and other resources are provided upon removing access to DISC-MA.

Participants can refuse and withdraw from participation at any time. If they withdraw consent from the study, they will no longer have access to the study treatment.

#### 8.1.3 Benefits

When evaluating the risks and benefits of the proposed study, it is believed that risks are relatively minimal when compared to the potential benefits that subjects are likely to receive. The benefits of engaging with DISC-MA include potentially improving mood (anxiety, stress, and/or depression), acquiring practical psychotherapeutic skills (from cognitive behavioral therapy, dialectical behavior therapy, and mindfulness), and receiving psychoeducation about mental health.

Participants who improve mood may derive additional benefits should said mood improvements be associated with other psychological improvements such as interpersonal or occupational functioning. Study of the effectiveness of this intervention will also benefit society more generally by providing data on the utility of Woebot.

#### **8.2 Adverse Events**

#### 8.2.1 Definitions

Adverse Event (AE): An AE is any unanticipated medical occurrence in a clinical study participant using an investigational product or from study procedures that does not necessarily have a causal relationship with this product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of an investigational product, whether or not related to the investigational product.

Serious Adverse Event (SAE): An SAE is any AE that meets any of the following criteria:

- Results in *death*
- Is life-threatening
- Requires inpatient *hospitalization* or prolongation of existing hospitalization
- Results in persistent or significant disability/incapacity
- Is a congenital anomaly/birth defect
- Is an *important medical event* that may not result in death, be life-threatening, or require
  hospitalization may be considered a serious adverse event when, based upon appropriate
  medical judgment, they may jeopardize the patient or subject and may require medical or
  surgical intervention to prevent one of the outcomes listed above.

<u>Unanticipated Problem (UAP):</u> A UAP is an incident, experience, or outcome that meets all of the following criteria:

• Unexpected in nature, severity, or frequency (i.e., not described in study-related documents such as the IRB- or IEC-approved protocol or consent form)

- Related or possibly related to participation in the research (i.e., possibly related means there is a
  reasonable possibility that the incident experience or outcome may have been caused by the
  procedures involved in the research)
- Suggests that the research places subjects or others at greater risk of harm (including physical, psychological, economic, or social harm)

An individual AE observed during the conduct of a study may be considered an unanticipated study problem involving risk to human subjects, and reported to the IRB, only if it is unexpected, serious, and would have implications for the conduct of the study (e.g., requiring a significant and, usually, safety-related change in the protocol such as revising the inclusion/exclusion criteria or including a new monitoring requirement or informed consent). Investigators should report possible UAP to the Sponsor and the Sponsor will make a determination for the UAP in the context of the study and any change to the study.

Adverse Device Effect (ADE): Any adverse event related to the use of an investigational medical device. This includes any adverse event resulting from insufficiencies or inadequacies in the instructions for use, the deployment, the implantation, the installation, the operation, or any malfunction of the investigational medical device. This also includes any event that is a result of a use error or intentional misuse.

<u>Unanticipated Adverse Device Effect (UADE)</u>: Any serious adverse effect on the health or safety, or any life-threatening problem or death caused by or associated with a device which was not previously identified in nature, severity or degree of incidence in the protocol, Instructions for Use, Summary of Previous Studies Document, or other sources of information for the investigational product. Additionally, a UADE is any other unanticipated serious problem associated with the investigational device that relates to the rights, safety, or welfare of subjects.

UADEs will include events meeting either A or B as stated below:

A. Events meeting ALL of the following criteria:

- Not included in the list of Anticipated Events (refer to protocol section 8.2.2)
- Related (possibly, probably, or definitely) to the investigational device per the site principal investigator
- Serious (meets any of the SAE criteria)

B. Any other unanticipated serious problem associated with the investigational device that relates to the rights, safety, or welfare of participants.

<u>Device Deficiencies:</u> Inadequacy of a medical device related to its identity, quality, durability, reliability, safety or performance, such as malfunction, misuse or use error and inadequate labeling. The reporting of a Device Deficiency is a Product Complaint.

<u>Product Complaints:</u> Any written, electronic, or oral communication that alleges deficiencies related to the identity, quality, durability, reliability, safety, effectiveness, or performance of a device after it is released for distribution.

#### **8.2.2 Previously Noted Adverse Device Effects**

Any ADE that is not identified in nature, severity, or is not listed below is considered unanticipated:

- Temporary upset may occur as a result of discontinued access to DISC-MA at the end of the study.
- Given that the study involves use of a smartphone application, there is the small possibility of unintended application outages.

#### **8.3** Assessment of Adverse Events

The investigator will be alert to any complaints or adverse reactions that arise and will take appropriate steps to Reduce the impact of any event . Existing disclaimers that DISC-MA is not intended for crisis management will be presented in the ICF and at onboarding. AEs may be received/identified via:

- 1) Spontaneous participant self reports communicated outside of the app
- 2) Solicited participant self reports collected via the Week 2 and Week 4 survey
- 3) Upon review of select conversations/transcripts with Woebot

Upon learning of a potential safety event, all relevant trial data will be compiled by a designated member of the study team and shared with the investigator. All events which meet criteria for an AE/SAE/UAP/UADE/Device Deficiency will be recorded by the PI or designee on the appropriate electronic Case Report Form (eCRF) and will follow a predetermined safety protocol as outlined in a Safety Management Plan (SMP).

#### 8.3.1 Time Frame

Collection of AEs and SAEs will begin at ICF signature, and will continue through EOS at Week 4. Identification of any collected AEs/SAEs from transcript or LDP reviews is anticipated to be completed no earlier than 1 month following the last patient visit and no longer than 4 months from the last patient visit or until all data has been monitored and query cleaned.

#### 8.3.2 AE Severity

If possible, investigators should report event terms that reflect a single, unifying diagnosis rather than individual signs or symptoms (e.g., "influenza" instead of "coughing, body aches, fever;" and "anemia" rather than "low hemoglobin"). A corresponding severity grading is to be performed by the investigator based on his/her best medical judgment as follows:

- Mild (Grade 1): asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated
- Moderate (Grade 2): minimal, local, or noninvasive intervention indicated; limited age-appropriate instrumental activities of daily living (ADL)

• **Severe (Grade 3):** medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; or limiting self-care ADL

- Life-threatening (Grade 4): life-threatening consequences; urgent intervention indicated
- Fatal (Grade 5): death related to an AE

#### 8.3.3 AE Causality

An event's relatedness to the investigational device will be determined by the Principal Investigator and classified under the following causality ratings:

- Non-related: There is no evidence of any causal relationship.
- **Related:** There is clear evidence of a casual relationship between the device and event; all other explanations have been ruled out.

#### 8.3.3 AE Outcomes

The Investigator should document the outcome of AE and SAEs as:

- Resolved
- Resolved with sequelae / chronic condition, no resolution expected
- Ongoing
- Death
- Ongoing at time of death
- Unknown

#### 8.4 Documenting and Reporting AE and SAEs

Designated members of the study team will report any identified potential safety events to the investigator within one business day from awareness. The investigator should seek to obtain information required to make a determination of causality and must assess the relationship of the event to the study device and complete the AE/SAE eCRF. Relevant follow up information should be updated as collected.

Any event that the Sponsor-Investigator determines is/are reportable to the IRB will be reported within 5 working days from making that determination. If it should be determined that an event presents an unreasonable risk to all participants, the study or parts of the study presenting that risk will be terminated as soon as possible.

## 8.5 Safety Monitoring

## 8.5.1 Safety Procedures At Screening

At screening, s tudy participants will be asked to self-report on recent suicidal thoughts including current suicidal ideation with plan and/or intent as well as attempts in the past 12 months. Responses are not monitored in real time. Participants who endorse having a current suicidal plan or intent or an attempt in the past 12 months will be excluded from the study. Participants will be notified that:

• They may benefit from a level of care beyond the scope of the study and investigational treatment.

- They should call 9-1-1 or go to their local emergency room and reach out to someone they trust and can help them stay safe if they feel they are in crisis or in need of medical attention.
- Will be electronically provided with a list of resources.

Participants who endorse <u>current</u> suicidal ideation with a plan <u>or</u> intent will also be notified that a member of the study team will attempt to follow-up with them. Three attempts will be made by the Study PI to contact participants by phone and/or email. The study team will make every effort to follow-up with the participant as soon as possible and no more than 3 business days following the initial report.

#### **8.5.2 Unscheduled Visits**

Study participants are able to initiate contact with the study team at anytime throughout the duration of the study. If the contact is attributable to safety reasons or if the study team learns about a suspected safety event at any time, then an Unscheduled Visit would ensue, wherein the qualified study personnel would attempt to follow-up with the participant, and if it is determined that they are in immediate risk for hurting themselves or others, appropriate steps would be taken as outlined in the study specific Safety Management Plan (SMP).

#### **8.5.3 Safety Event Solicited Self-Report Survey**

Study participants will be asked to self-report on potential safety events at the Week 2 and Week 4 timepoints. Questions will explicitly ask about changes in the past two weeks to their (1)medication and/or therapy, (2) mental and/or physical health, and (3) any new thoughts about ending their life including new intent/plan/or attempts. Information gathered through this survey will be used to inform the need for follow-up, AEs/SAEs/UAPs/UADEs/Device Deficiencies/UADE determination, and resolution.

#### 8.5.4 Language Detection Protocol (LDP)

In addition to the onboarding screens re-stating that Woebot is not a crisis service, DISC-MA has a Language Detection Protocol (LDP), developed by Woebot Health. The purpose of the LDP is to detect potentially concerning topics within participant-input free-text and will be enacted for all participants in the study . Upon detection of any concerning topics, LDP initiates a conversation to remind the participant of the application's limitations of services and offer a resource list which includes readily accessible support channels. If a possible mention of concerning topics is detected, the participant is reminded of the limitations of services (which they will have already seen in both the informed consent and well as Woebot's onboarding screens) as well as offered a list of external-to-application resources, specifically contact information, that have been curated in consultation with suicide prevention experts. This resource list includes emergency contact phone numbers, and suicide ideation and domestic violence hotline information.



Woebot Health Version 1.1

W-DISC-002 18/MAR/2024





# 8.6 Safety Assessment Committee (SAC)

The SAC is the formal WH committee charged with responsibility for the review and evaluation of previous as well as accumulating data from clinical studies of WH devices, to assess safety, perform signal confirmation and risk assessment, assess the risk-benefit associated with study continuation, efficacy and other trial conduct issues such as scientific merit, and to develop recommendations so as to ensure safety across studies and minimize risk for subjects. The SAC members will include the following individuals:

- 1. Independent Medical Safety Expert, who will serve as the SAC Chair;
- 2. A Clinical Development Lead;
- 3. a Medical Lead;
- 4. a Regulatory Lead;
- 5. a Device Vigilance Lead

Validated, accurate and interpretable data are to be provided to the SAC, as requested. Data files to be used for SAC analyses will undergo established data review/QC procedures to the extent possible and critical fields will be identified. The Sponsor must ensure that data is of sufficient quality to support the performance of safety surveillance and confirm the assessment of causality associated with the event(s), the associated WH application and confirmation of reportability.

The SAC will determine whether any missing data will significantly impact the safety assessment and will direct the necessary actions to address missing data.

# 8.7 Quality Control and Quality Assurance

The Sponsor maintains a robust Quality Management System (QMS) that includes all activities involved in quality assurance and quality control per 21 CFR 820, to ensure compliance with written SOPs as well as applicable global/local GCP regulations and ICH Guidelines.

Audits of investigator sites, vendors, and Sponsor systems are performed by auditors, independent from those involved in conducting, monitoring, or performing quality control of the clinical trial. The clinical audit process uses a knowledge/risk-based approach.

Audits are conducted to assess 21 CFR 820 and GCP compliance with global and local regulatory requirements, protocols and internal SOPs and are performed according to specified Sponsor processes.

# 9. Statistical Analysis

# 9.1 General Methodology

Given the exploratory nature of this study, and its hypothesis-generating purpose, analyses will be descriptive in nature and will not include significance testing. Descriptive statistics for all endpoints will be reported for the full sample. All continuous variables will be tested for normality using a skewness cutoff of 1.00. For continuous variables, means and standard deviations will be reported if the data are normally distributed; for non-normal data, medians and interquartile ranges will be reported. Frequencies and percentages will be reported for categorical variables. The amount of missing data will be summarized. Where applicable, bivariate comparisons will be conducted using chi-squared tests, Fisher exact test, t-tests, one-way ANOVA, Person's correlation, and Spearman's correlation. However, no hypothesis testing will be completed, and only effect sizes and 95% confidence intervals will be provided where applicable. For departures from normality, the appropriate non-parametric method will be applied.

#### 9.2 Analysis Sets

Primary analyses will be completed on two sets of data - the full intent-to-treat (ITT) sample of anyone randomized with available survey data, as well as a per-protocol (PP) sample (i.e., registered for app, completed all assessment timepoints, no protocol deviations, etc).

# 9.3 Sample Size Determination

No formal sample size calculations were performed due to the exploratory nature of this study; however, N=200 was targeted to allow for a large enough sample to sufficiently explore potency and precision patterns, and certain health equity outcomes (depending on sample diversity and attrition).

## **10. Statistical Methods**

## **10.1 Primary Endpoint**

#### 10.1.1 Aim

Describe therapeutic alliance with Woebot at week 1 and week 4 of the intervention.

# 10.1.2 Hypothesis

Understanding aspects of the working alliance between users and Woebot at both the beginning and end of treatment will provide hypotheses for the future development of precision interventions.

#### 10.1.3 Endpoints

Therapeutic alliance will be measured by the Working Alliance Inventory (WAI) total scale score at week 1 and WAI total scale score at week 4.

#### 10.1.4 Analysis Plan

Descriptive statistics will be used to describe therapeutic alliance at week 1 and week 4 of the intervention. Descriptive statistics will also summarize socio-demographic characteristics of the sample.



# **10.3 Safety Endpoints**

#### 10.3.1 Aims and Endpoints

The safety profile of DISC-MA will be investigated as an exploratory aim and measured through:



- Frequency of AE/SAE/UADEs
  - Spontaneous participant report of safety events that are determined to be an AE/SAE/UADE
  - Direct participant self-report of safety events at the Week 2 and Week 4 survey that are determined to be an AE/SAE/UADE
  - Transcript reviews that detect safety events and are determined to be an AE/SAE/UADE

#### 10.3.2 Analysis of Safety

To observe and describe upon the utilization and outcomes of the safety procedures utilized within this study (e.g., AE/SAEs and device relatedness). For each safety endpoint, n(%) will be reported.

## **10.4 Demographic and Baseline Characteristics**

Demographic and baseline characteristics will be summarized for the full sample. Continuous variables will be summarized using tables of descriptive statistics, with normally distributed variables summarized by mean and standard deviation and non-normal data summarized by median and interquartile range (IQR). Categorical and ordinal variables will be described using frequencies and percentages.

#### **10.5** Handling of Missing Values

Frequencies of missing values will be indicated in all descriptive tables, and no imputation or other statistical manipulation will be used for missing values.

#### 11. Ethics and Responsibilities

#### **11.1 Good Clinical Practice**

This study will be conducted in accordance with the Note for Guidance on GCP ICH Harmonised Tripartite Guideline E6 (R1)/Integrated Addendum E6 (R2); US FDA Code of Federal Regulation (CFR) (Title 21 Parts 50, 56, 312); the general guidelines indicated in the Declaration of Helsinki; and all applicable regulatory requirements.

#### 11.2 Institutional Review Board

The final study protocol, including the final version of the ICF, must be approved, or given a favorable opinion in writing from the IRBs as appropriate. A written approval from the IRB is required for any study protocol amendment(s), ICF updates, participant recruitment procedures (e.g., advertisements), and any written information to be provided to participants and a statement from IRB to ensure compliance with GCP requirements (if applicable). The investigator is required to sign a protocol signature page confirming their agreement to conduct the study in accordance with the document and all of the instructions and procedures found in this protocol and to give access to all relevant data and records to Sponsor monitors, auditors, Sponsor Quality assurance representatives, designated agents of Sponsor, IRBs, and regulatory authorities as required.

The IRB approval must identify the protocol version as well as the documents reviewed. Any amendments to the protocol will require IRB approval before the implementation of the changes made to the study, except for changes necessary to eliminate an immediate hazard to the study participants.

The investigator will be responsible for the following:

- Providing written summaries of the status of the study to the IRB annually or more frequently in accordance with the requirements, policies, and procedures established by the IRB
- Notifying the IRB of SAEs or other significant safety findings as required by IRB procedures
- Providing oversight of the conduct of the study at the site and adherence to the requirements of all applicable regulations
- Promptly reporting deviations from, or changes to, the protocol to eliminate immediate hazards to the study participants

#### 11.3 Informed Consent

In obtaining and documenting consent via an Electronic Informed Consent Form (eICF), the investigator should comply with the applicable regulatory requirement(s) and should adhere to GCP and to the ethical principles that have their origin in the Declaration of Helsinki. Prior to the beginning of the study, the investigator should have the IRB's written approval/favorable opinion of the eICF and any other pertinent information to be provided to participants.

- Following completion of pre-screening, participants will be provided with a link to the eICF where they will have the opportunity to independently review and determine whether they are interested in participating.
- Participants will be provided with contact information for the study team whom they can reach out to with any questions prior to signing the eICF.
- Participants are informed that their participation is voluntary, and consent can be withdrawn at any point.
- Participants will be required to sign a statement of informed consent that meets the requirements of US FDA CFR Title 21 Part 50, local regulations, ICH guidelines, HIPAA requirements in the US, and the IRB or study site.

• Prior to a participant's participation in the study, the eICF should be signed and personally dated by the participant.

- An electronic copy of the signed eICF will be retained by the study team.
- A copy of the eICF and any other pertinent information must be provided to the participant.
- If the eICF is revised, the revised eICF must have received the IRB's approval/favorable opinion in advance of its use. Participants must be informed of the changes to the eICF and must re-consent to the most current version during their participation in the study if the IRB confirms the change requires re-consent. The participant should be informed in a timely manner if new information becomes available that may be relevant to the participant's willingness to continue participation in the study. The communication of this information should be documented.

# 12. Records Management

All clinical study information should be recorded, handled, and stored in a way that allows its accurate reporting, interpretation, and verification. This principle applies to all records referenced in this protocol, irrespective of the type of media used. All records will be collected and maintained via secure and approved online platforms.

Details regarding eCRF access and handling are detailed in the "Electronic Case Report Form Completion and Data Management" section.

Any contact with the participant via telephone or other means that provides significant clinical information is to be documented and maintained as part of the study record. Information from the study records and other source documents is to be promptly entered into the appropriate section of the eCRF.

Changes to information in the study record and other source documents will be electronically tracked. If the reason for the change is not apparent, a brief explanation for the change is to be written adjacent to the change.

The lead biostatician will write a data management plan, which will be finalized prior to performing any data validation.

#### **12.1 Source Documentation**

Source documents will be collected electronically. Source documents contain the results of original observations and activities of this research study. They are the original records in which raw data are first recorded. Source documents include, but are not limited to screening logs, consent forms, and recorded data from automated instruments.

The investigator/study personnel should maintain adequate and accurate source documents and study records that include all pertinent observations on each of the study participants. Source data should be attributable, legible, contemporaneous, original, accurate, and complete. Changes to source data should be traceable, should not obscure the original entry, and should be explained if necessary (e.g., via an audit trail).

All source documents from this study are to be maintained by the investigator and made available for inspection by authorized persons. The investigator will provide direct access to source documents/data for study-related monitoring, audits, IRB review, and regulatory inspections. The Sponsor-Investigator should verify that each participant has consented, in writing, to direct access to his/her original study records for study-related monitoring, audit, IRB review, and regulatory inspection.

#### 12.2 Case Report Form Completion and Data Management

Access to the eCRF will be strictly password protected and limited to personnel directly participating in the study. Data should be entered into the eCRF completely by authorized site personnel (e.g., investigators and the study coordinator). The eCRF must be completed as soon as possible (no later than 5 business days) after any participant evaluation or communication. Changes to the eCRF will be electronically tracked.

Data will be entered/loaded into a validated online platform. Computerized data cleaning checks will be used in addition to manual review to check for discrepancies and to ensure consistency of the data.

# 12.3 Study Files and Record Retention

All data derived from the study will remain the property of the Sponsor-Investigator. The Sponsor-Investigator assumes accountability for actions delegated to other individuals (e.g., CRO, other study personnel).

Records must be retained in accordance with the current ICH Guidelines on GCP. All essential study documents, including records of participants, source documents, and eCRFs must be kept on file.

Essential documents should be retained until at least 2 years after the last approval of a marketing application in an ICH region and until there are no pending or contemplated marketing applications in an ICH region, or until at least 2 years have elapsed since the formal discontinuation of clinical development of the investigational product. However, essential documents may be retained for a longer period if required by the applicable regulatory requirements or by agreement with the Sponsor. The Sponsor is responsible for informing the investigator when these documents need no longer be retained.

The investigator is not to dispose of any records relevant to this study without written permission from the Sponsor and is to provide the Sponsor the opportunity to collect such records. The investigator shall take responsibility for maintaining adequate and accurate hard copy source documents, if utilized, of all observations and data generated during this study. Such documentation is subject to inspection by the Sponsor, its representatives, and regulatory authorities.

If an investigator moves, withdraws from a study, or retires, the responsibility for maintaining the records may be transferred to another person who will accept responsibility. Notice of transfer must be made to and agreed by the Sponsor.

# 13. Auditing and Monitoring

Quality control will occur at each stage of data handling to ensure that all data are reliable and have been processed correctly. The Sponsor-Investigator should ensure oversight of any study-related duties

and functions carried out on its behalf, including study-related duties and functions that are subcontracted to another party by the Sponsor's contracted vendors or other study personnel.

The eCRFs should be completed in a timely manner and on an ongoing basis to allow regular review by the study monitor or designee.

Details describing the strategy, responsibilities, and requirements of the study monitoring are provided in the study monitoring plan.

The purpose of an audit is to assess whether ethics, regulatory, and quality requirements are being fulfilled. The Sponsor or its representative may conduct audits including, but not limited to, presence of required documents, the informed consent process, and comparison of eCRFs with source documents. Government regulatory authorities may also conduct an inspection during or after the study. All study records must be available for audit. The Sponsor-Investigator must agree to participate with audits conducted at a convenient time in a reasonable manner.

#### 13.1 Protocol Adherence and Deviations

The investigator and study personnel should conduct the study in compliance with the protocol and should use continuous vigilance to identify and report protocol deviations.

A protocol deviation is any change, divergence, or departure from the study design or procedures defined in the protocol that may be on the part of the investigator, site personnel, or the participant.

Protocol violations are a subset of protocol deviations that may significantly impact the completeness, accuracy, and/or reliability of the study data or that may significantly affect a participant's rights, safety, or well-being. For example, important protocol deviations may include enrolling participants in violation of key eligibility criteria designed to ensure a specific participant population or failing to collect data necessary to interpret primary endpoints, as this may compromise the scientific value of the study.

The investigator should not implement any deviation from the protocol without agreement from the Sponsor and prior review and approval from the IRB of an amendment, except where necessary to eliminate an immediate hazard to a study participant, or when the change involves only logistical or administrative aspects of the study, such as a change in a monitor or telephone number.

In the event of an important protocol deviation, the investigator will report the deviation to the SAC, as described in the SMP, and will come to an agreement as to whether the participant should be withdrawn from the study due to the important protocol deviation.

## 14. Amendments

Protocol modifications, except those intended to reduce immediate risk to study participants, may be made only by the Sponsor. A protocol change intended to eliminate an apparent immediate hazard to participants should be implemented immediately.

Any permanent change to the protocol must be handled as a protocol amendment. The written amendment must be submitted to the IRB, and the investigator must await approval before

implementing the changes. The Sponsor will submit protocol amendments to the appropriate regulatory authorities for approval.

The current version of the ICF will require similar modification if the IRB, investigator, and/or Sponsor, judge the amendment to the protocol to substantially change the study design and/or increase the potential risk to the participant and/or impact the participant's involvement as a study participant. In such cases, the ICF will be renewed for enrolled participants before their continued participation in the study.

# 15. Study Start and Termination

The study start date is the date on which the first participant provides informed consent.

The end of the study is defined as the last participant's last assessment.

Both the Sponsor and the investigator reserve the right to terminate the study or the participation in the study at an investigator's site at any time. In terminating the study, the Sponsor and the investigator will assure that adequate consideration is given to the protection of the participants' interests.

If the study is prematurely terminated or suspended for any reason, the Sponsor-Investigator or designated study personnel should promptly inform the study participants and should assure appropriate therapy and follow-up for the participants. Where required by the applicable regulatory requirements, the IRB, and other entities involved in the study should be informed promptly and be provided with a detailed written explanation of the termination or suspension.

#### **16. Confidentiality**

All information generated in this study is considered highly confidential and must not be disclosed to any person or entity not directly involved with the study unless prior written consent is gained from the Sponsor. However, authorized regulatory officials, IRB personnel, the Sponsor and its authorized representatives are allowed full access to the records.

All study participants must be informed that their personal study-related data will be used by the Sponsor in accordance with local data protection law. The level of disclosure must also be explained to the participant, who will be required to give consent for their data to be used as described in the ICF. Participants must be informed that their medical records may be examined by auditors or other authorized personnel appointed by the Sponsor, by appropriate IRB members, and by inspectors from regulatory authorities.

Identification of participants and eCRFs shall be by unique participant identification numbers (such as screening or randomization number) only. All personal identifiers according to applicable regulations (e.g., name, phone number) must be redacted permanently by the site personnel and replaced with the participant 's unique identification number in all records and data before transfer to the Sponsor (or designee).

All personal details will be treated as confidential by the investigator and study team members.

Woebot Health Version 1.1

W-DISC-002 18/MAR/2024

#### 17. References

1. Center for Devices and Radiological Health. Precision Medicine. U.S. Food & Drug Administration (FDA). Published August 18, 2023. Accessed December 21, 2023. https://www.fda.gov/medical-devices/in-vitro-diagnostics/precision-medicine

- 2. Fernandes BS, Williams LM, Steiner J, Leboyer M, Carvalho AF, Berk M. The new field of 'precision psychiatry.' *BMC Med*. 2017;15(1):80. doi:10.1186/s12916-017-0849-x
- 3. Kroenke K, Strine TW, Spitzer RL, Williams JBW, Berry JT, Mokdad AH. The PHQ-8 as a measure of current depression in the general population. *J Affect Disord*. 2009;114(1-3):163-173. doi:10.1016/j.jad.2008.06.026
- 4. Spitzer RL, Kroenke K, Williams JBW, Löwe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. *Arch Intern Med.* 2006;166(10):1092-1097. doi:10.1001/archinte.166.10.1092
- 5. Munder T, Wilmers F, Leonhart R, Linster HW, Barth J. Working Alliance Inventory-Short Revised (WAI-SR): psychometric properties in outpatients and inpatients. *Clin Psychol Psychother*. 2010;17(3):231-239. doi:10.1002/cpp.658
- 6. Dennis J, Vander Wal J. The Cognitive Flexibility Inventory: Instrument Development and Estimates of Reliability and Validity. *Cogn Ther Res.* 2010;34:241-253. doi:10.1007/s10608-009-9276-4
- 7. Kaufman E, Xia M, Fosco G, Yaptangco M, Skidmore C, Crowell S. The Difficulties in Emotion Regulation Scale Short Form (DERS-SF): Validation and Replication in Adolescent and Adult Samples. *J Psychopathol Behav Assess.* 2016;38. doi:10.1007/s10862-015-9529-3
- 8. Gard D, Germans Gard M, Kring A, John O. Anticipatory and consummatory components of the experience of pleasure: a scale development study. *J Res Personal*. 2006;40:1086-1102. doi:10.1016/j.jrp.2005.11.001
- 9. Cyranowski JM, Zill N, Bode R, et al. Assessing social support, companionship, and distress: National Institute of Health (NIH) Toolbox Adult Social Relationship Scales. *Health Psychol*. 2013;32(3):293-301. doi:10.1037/a0028586
- 10. Terides MD, Dear BF, Karin E, et al. The frequency of actions and thoughts scale: development and psychometric validation of a measure of adaptive behaviours and cognitions. *Cogn Behav Ther*. 2016;45(3):196-216. doi:10.1080/16506073.2016.1149876
- 11. Centers for Medicare and Medicaid Services, Billioux A, Verlander K, et al. Standardized Screening for Health-Related Social Needs in Clinical Settings: The Accountable Health Communities Screening Tool. *NAM Perspect*. 2017;7(5). doi:10.31478/201705b